CLINICAL TRIAL: NCT01766401
Title: A Double-Blind, Placebo-Controlled, Flexible-Dose Study of Vilazadone in Patients With Generalized Anxiety Disorder
Brief Title: Safety, Efficacy and Tolerability of Vilazodone in Patients With Generalized Anxiety Disorder
Acronym: VLZ-MD-06
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLZ-MD-06
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; GAD
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Administration, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo tablets, oral administration
  Interventions: Drug: Placebo
- Vilazadone (Experimental): Vilazadone tablets, oral administration
  Interventions: Drug: Vilazadone

INTERVENTIONS:
Drug: Placebo
  Other Names: Dose-matched placebo tablets, oral administration, once per day
  Arms: Placebo
Drug: Vilazadone — Viibryd
  Other Names: Vilazadone once per day, 20 mg dose, oral administration or Vilazadone once per day, 40 mg dose, oral administration.
  Arms: Vilazadone

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of vilazodone relative to placebo in the treatment of generalized anxiety disorder (GAD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18 - 70 Years of age
* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for Generalized Anxiety Disorder (GAD)
* Minimum score of 20 on the Hamilton Rating Scale for Anxiety (HAM-A)

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control
* Patients with a history of meeting DSM-IV-TR criteria for:

  * any manic, hypomanic or mixed episode, including bipolar disorder and substance-induced manic, hypomanic, or mixed episode;
  * any depressive episode with psychotic or catatonic features;
  * panic disorder with or without agoraphobia;
  * obsessive-compulsive disorder;
  * Schizophrenia, schizoaffective, or other psychotic disorder;
  * bulimia or anorexia nervosa;
  * presence of borderline personality disorder or antisocial personality disorder;
  * mental retardation, dementia, amnesia, or other cognitive disorders
* Patients who are considered a suicide risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2014-01-29 (Actual); Study Completion 2014-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Forero, MA, Study Director — Forest Laboratories
Locations (30):
- United States (30):
  - Forest Investigative Site 022, Arcadia, California
  - Forest Investigative Site 023, Beverly Hills, California
  - Forest Investigative Site 010, Encino, California
  - Forest Investigative Site 025, Newport Beach, California
  - Forest Investigative Site 004, Redlands, California
  - Forest Investigative Site 007, Sherman Oaks, California
  - Forest Investigative Site 016, Temecula, California
  - Forest Investigative Site 012, Upland, California
  - Forest Investigative Site 017, Coral Springs, Florida
  - Forest Investigative Site 028, Fort Myers, Florida
  - Forest Investigative Site 002, Jacksonville, Florida
  - Forest Investigative Site 020, Leesburg, Florida
  - Forest Investigative Site 024, Miami, Florida
  - Forest Investigative Site 001, Orlando, Florida
  - Forest Investigative Site 026, Indianapolis, Indiana
  - Forest Investigative Site 029, Shreveport, Louisiana
  - Forest Investigative Site 019, Las Vegas, Nevada
  - Forest Investigative Site 003, Canton, Ohio
  - Forest Investigative Site 031, Columbus, Ohio
  - Forest Investigative Site 021, Mason, Ohio
  - Forest Investigative Site 030, Oklahoma City, Oklahoma
  - Forest Investigative Site 005, Salem, Oregon
  - Forest Investigative Site 014, Allentown, Pennsylvania
  - Forest Investigative Site 015, Philadelphia, Pennsylvania
  - Forest Investigative Site 027, Lincoln, Rhode Island
  - Forest Investigative Site 006, Memphis, Tennessee
  - Forest Investigative Site 008, Houston, Texas
  - Forest Investigative Site 018, Houston, Texas
  - Forest Investigative Site 011, Murray, Utah
  - Forest Investigative Site 013, Woodstock, Vermont

REFERENCES:
- [Derived] Khan A, Durgam S, Tang X, Ruth A, Mathews M, Gommoll CP. Post Hoc Analyses of Anxiety Measures in Adult Patients With Generalized Anxiety Disorder Treated With Vilazodone. Prim Care Companion CNS Disord. 2016 Apr 28;18(2):10.4088/PCC.15m01904. doi: 10.4088/PCC.15m01904. eCollection 2016. PMID 27486544
- [Derived] Gommoll C, Forero G, Mathews M, Nunez R, Tang X, Durgam S, Sambunaris A. Vilazodone in patients with generalized anxiety disorder: a double-blind, randomized, placebo-controlled, flexible-dose study. Int Clin Psychopharmacol. 2015 Nov;30(6):297-306. doi: 10.1097/YIC.0000000000000096. PMID 26291335

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Dose-matched placebo tablets, oral administration, once per day
- Vilazadone: Vilazadone once per day, 20 mg dose, oral administration or Vilazadone once per day, 40 mg dose, oral administration.
Period: Overall Study
Arm/Group | Placebo | Vilazadone
Started | 198 | 200
Completed | 161 | 144
Not Completed | 37 | 56
Not completed — Adverse Event | 7 | 22
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 3 | 8
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Lost to Follow-up | 10 | 11
Not completed — Pregnancy | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilazadone | Total
Number analyzed (Participants) | 198 | 200 | 398
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (13.0) | 40.5 (13.2) | 40.3 (13.1)
Age, Customized [Number; unit: Participants]
  < 20 | 3 | 5 | 8
  20-29 | 48 | 50 | 98
  30-39 | 51 | 45 | 96
  40-49 | 41 | 40 | 81
  50-59 | 37 | 45 | 82
  ≥ 60 | 18 | 15 | 33
Sex/Gender, Customized [Number; unit: Participants]
  Male | 67 | 55 | 122
  Female | 131 | 145 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 46 | 83
  Not Hispanic or Latino | 161 | 154 | 315
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 160 | 164 | 324
  Black or African American | 32 | 23 | 55
  Asian | 3 | 9 | 12
  American Indian or Alaska Native | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline in the Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
Time Frame: Baseline to Week 8
Population: The Intent-to-Treat (ITT) Population consisted of all patients in the Safety Population who had at least 1 postbaseline assessment of the HAM-A.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Placebo | Vilazadone
Number analyzed (Participants) | 197 | 198
Score on Scale | 14.9 (7.37) | 13.5 (7.41)
Statistical Analysis 1: Comparison: Placebo vs Vilazadone; Test type: Superiority; p = 0.0438, MMRM; Least Squares Mean Difference = -1.50, 95% CI 2-sided [-2.96 to -0.04]

2. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe).
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Placebo | Vilazadone
Number analyzed (Participants) | 197 | 198
Score on Scale | 10.1 (6.58) | 7.8 (6.91)
Statistical Analysis 1: Comparison: Placebo vs Vilazadone; Test type: Superiority; p = 0.0868, MMRM; Least Squares Mean Difference = -1.41, 95% CI 2-sided [-3.02 to 0.20]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until week 8.
Description: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Vilazadone
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/200
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/200
Other Adverse Events (participants affected / at risk) | 75/198 | 130/200
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=198) | Vilazadone (N=200)
Nausea (Gastrointestinal disorders) | 19 | 63
Diarrhoea (Gastrointestinal disorders) | 24 | 62
Vomiting (Gastrointestinal disorders) | 2 | 13/198
Dry mouth (Gastrointestinal disorders) | 10 | 11
Upper respiratory tract infection (Infections and infestations) | 10 | 9
Dizziness (Nervous system disorders) | 14 | 15
Headache (Nervous system disorders) | 21 | 15
Somnolence (Nervous system disorders) | 6 | 12
Abnormal dreams (Psychiatric disorders) | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the PI will be subject to mutual agreement between the PI and Forest Research Institute, Inc.